CLINICAL TRIAL: NCT00247299
Title: Evaluation and Optimization of the Technical and Clinical Performance of the Lumenis ONE Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Lumenis Be Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: danaCTIL; danaCTIL
Record Dates: First submitted 2005-10-30; First posted 2005-11-01 (Estimated); Last update posted 2005-11-01 (Estimated); Status verified 2005-10

CONDITIONS: Telangiectases; Port Wine Stain
Keywords: Vascular lesions; Intense pulse light; phototermolysis; wavelength; filters; non coherent
MeSH Terms: conditions — Telangiectasis; Port-Wine Stain

INTERVENTIONS:
Device: IPL Quantum Product manufactured by Luminis Ltd.

SUMMARY:
The Intense Pulsed Light (IPL) technology, by selective phototermolysis, is used for eliminating, among other application, benign vascular lesions and unwanted leg veins. Light energy heats the deeper structures of the skin. IPL devices provide a broad wavelength spectrum of 515 to 1200 nm and fluence from 10 to 40 J/cm at o.5-1 Hz.The light is focused by a reflector and then transmitted through various filters that cut off the lower wavelength range of the emitted light; therefore, only those wavelengths longer than these of the filters are transmitted.

objectives:

1. evaluate and optimize the clinical performance of the Luminis ONE platform for each of the aforementioned clinical applications.
2. Reconfirm the parameter settings for each of the aforementioned clinical applications.
3. Confirm the user friendly design of the device, in aspects of software (user interface) and various technical operational features.

DETAILED DESCRIPTION:
Background:

The Intense Pulsed Light (IPL) technology, by selective phototermolysis, is used for eliminating, among other application, benign vascular lesions and unwanted leg veins. Light energy heats the deeper structures of the skin. IPL devices provide a broad wavelength spectrum of 515 to 1200 nm and fluence from 10 to 40 J/cm at o.5-1 Hz.The light is focused by a reflector and then transmitted through various filters that cut off the lower wavelength range of the emitted light; therefore, only those wavelegths longer than these of the filters are transmitted.

Material and Methods:

The luminis ONE medical system (Lumenis Ltd., Yokneam,Israel, and Pleasanton, CA, USA) incorporate the non coherent pulsed light head.

Vascular lesion such as Telangiectases, leg veins or PWS will be treated with the IPL, with the following filters :515,50,or 590.

Following every treatment the subjects will be asked how much pain was felt , using a score of 1-5.

Photographs will be taken before each treatments . Every subject will be treated 5 treatments , with 5+1 weeks interval. clearance or improvement will be evaluated by the physician at each visit,before the next treatment using the following scale:

1. No clearance
2. 0-25%
3. 25-50%
4. 50-75%
5. 75-100%

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects, presenting with at least one of the clinical indications mentioned above
* Willing and being able to comply with all visit and evaluation requirements
* Willing and being able to provide signed Informed Consent

Exclusion Criteria:

* A history of keloid scar formation or poor wound healing
* Wounded or tanned in area to be treated
* Pregnant or intending to become pregnant during the evaluation period
* Subjects with a bleeding disorder or who take anticoagulation medications
* Significant concurrent illnesses, such as diabetes, epilepsy, lupus or congestive heart failure
* Significant concurrent skin conditions affecting area to be treated
* Having a history of skin cancer or any other cancer in the area to be treated
* History of immunosuppressive disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-05

PRIMARY OUTCOMES:
Every subject will be treated 5 treatments , with 5+1 weeks interval.
clearance or improvement will be evaluated by the physician at each visit,before the next treatment using the following scale:
1. No clearance
2. 0-25%
3. 25-50%
4. 50-75%
5. 75-100%

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullmann, MD, Principal Investigator — Plastic Surgery Dept., Rambam Medical Center., Haifa,Israel
Locations (1):
- Plastic surgery dept., Rambam medical center, Haifa, Israel